CLINICAL TRIAL: NCT02398110
Title: Transvaginal NOTES Nephrectomy Versus Conventional Laparoscopic Nephrectomy: a Randomized Clinical Trial
Brief Title: Transvaginal NOTES Nephrectomy Versus Conventional Laparoscopic Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Gannan Medical University (Other)
Responsible Party: Principal Investigator, Xiaofeng Zou, professor, First Affiliated Hospital of Gannan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20121BBG70032
Record Dates: First submitted 2015-03-10; First posted 2015-03-25 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transvaginal NOTES nephrectomy (Experimental): A 5- and 10-mm trocar were placed at the right and left medial margin of umbilicus. A lengthened 10-mm trocar was placed through the vagina into the abdominal cavity
  Interventions: Procedure: transvaginal NOTES nephrectomy; Procedure: conventional laparoscopic nephrectomy
- conventional laparoscopic nephrectomy (Active Comparator): One 10-mm trocar was inserted at the midclavicular line 2 cm below the umbilicus, another 10-mm periumbilical trocar was placed for the camera, and a 5- or 10-mm trocar was placed 3 cm below the costal margin
  Interventions: Procedure: transvaginal NOTES nephrectomy; Procedure: conventional laparoscopic nephrectomy

INTERVENTIONS:
Procedure: transvaginal NOTES nephrectomy — A 5- and 10-mm trocar were placed at the right and left medial margin of umbilicus. A lengthened 10-mm trocar was placed through the vagina into the abdominal cavity
Procedure: conventional laparoscopic nephrectomy — One 10-mm trocar was inserted at the midclavicular line 2 cm below the umbilicus, another 10-mm periumbilical trocar was placed for the camera, and a 5- or 10-mm trocar was placed 3 cm below the costal margin

SUMMARY:
Recent reports have suggested that transvaginal NOTES nephrectomy is feasible, yet comparative studies are lacking. The aim of this study was to compare the surgical outcomes of transvaginal NOTES nephrectomy to conventional laparoscopic nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* indication for nephrectomy due to benign or malignant kidney disease,
* age between 18 and 65 years, and
* legal competence

Exclusion Criteria:

* emergency surgery,
* contraindications to laparoscopic surgery,
* class IV or V as defined by the American Society for Anesthesiologists (ASA),
* body mass index (BMI) of > 30 kg/m2,
* advanced TNM staging (≥ T3),
* history of major abdominal surgery,
* gravidity or breast-feeding, and
* no written informed consent signed

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain in motion (Pain Scores on the Visual Analog Scale (0-10) | at postoperative day 1
  Pain Scores on the Visual Analog Scale (0-10)

SECONDARY OUTCOMES:
Cosmetic assessment (Patient Scar Assessment Questionnaire) | > 3 months after surgery
  The cosmetic result was assessed using a Patient Scar Assessment Questionnaire and Scoring System (PSAQ)
Sexual function (Female Sexual Function Index) | Preoperatively, and 4, 8 and 12 months postoperatively
  Sexual function was evaluated according to the Female Sexual Function Index
Intraoperative complications (e.g. bleeding, organ-injury) | Evaluated at the operation day
  e.g. bleeding, organ-injury
Duration of the operation | at the operation day
  in minutes
Quality of life (SF-36) | on postoperative month 1
  measured with the
Postoperative complication (classified using the Clavien-Dindo system) | early (≤ 1 month), or late (>1 month)
  Early (≤ 1 month) and late (> 1 month) complications were classified using the Clavien-Dindo system

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi, China